CLINICAL TRIAL: NCT02163681
Title: MRI as a Means to Measure Lung Function: Non-Invasive Imaging in Neonates and Young Children
Brief Title: MRI for Non-Invasive Imaging in Neonates and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Xemed LLC (Industry)
Responsible Party: Principal Investigator, Y. Michael Shim, MD, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15720
Record Dates: First submitted 2014-06-10; First posted 2014-06-16 (Estimated); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Healthy; Cystic Fibrosis (CF); Asthma; Bronchopulmonary Dysplasia (BPD)
MeSH Terms: conditions — Cystic Fibrosis; Asthma; Bronchopulmonary Dysplasia

ARMS (1):
- Hyperpolarized Helium 3 MRI of the chest (Experimental): Using hyperpolarized helium-3 as an inhaled contrast agent for MRI, we will assess the lung ventilation.
  Interventions: Drug: Hyperpolarized Helium-3 MRI of the chest

INTERVENTIONS:
Drug: Hyperpolarized Helium-3 MRI of the chest — hyperpolarized helium-3 is an inhaled gaseous contrast agent for MRI and permits the acquisition of high quality imagined of lung ventilation.

SUMMARY:
The purpose of this study is to develop rapid MRI techniques for imaging the lung with hyperpolarized helium-3 gas as an inhaled contrast agent. These techniques will be piloted in adults and older children before testing them in younger children and infants. The purpose is to enable imaging of non-sedated infants by imaging so fast as to freeze motion.

DETAILED DESCRIPTION:
he purpose of this study is to further develop the techniques to permit the imaging of infant lungs with hyperpolarized helium-3 MRI including techniques for acquisition in free breathing infants and infants on a ventilator. We have developed fast imaging techniques and obtained proof-of-concept data in infants as young as 2 months old. Many pediatric lung diseases including CF, bronchopulmonary dysplasia (BPD) and asthma have their origins in infancy so it would be desirable to be able to image infants with hyperpolarized gas MRI. We focused on developing fast imaging techniques to, in essence, freeze lung motion in non-sedated infants. We feel the technique will be more widely adopted if clinically useful images can be obtained without sedating the infant. Some very rapid imaging techniques have been developed for conventional proton MRI for applications such as cardiac MRI that require very short acquisition time. We modified these techniques for use in hyperpolarized gas MRI and developed a technique that permits the acquisition of the entire lung volume of an infant in less than 1 second. These techniques would also be useful for imaging infants who are still on a ventilator with the hope of increasing our understanding of lung development and neonatal lung disease.

ELIGIBILITY:
Inclusion Criteria:

* MRI sequence development (n=40): Healthy subjects and patients with CF, BPD, or asthma will be used in the development of the rapid imaging techniques. These subjects will be age 4 months to 65 years old. Healthy subjects can have no history of chronic respiratory disease. The subjects with CF or asthma must have a physician diagnosis of their respective disease.
* Proof-of-Concept Study (n=30): Ten healthy infants,10 infants with CF, and 10 infants with BPD age 4-24 months will be imaged in the proof-of-concept study. Healthy infant must have had an uncomplicated term birth and have no history of chronic respiratory symptoms. The patients with CF must have a physician diagnosis of CF and be at their baseline clinical status on the day of imaging.

Exclusion Criteria:

* Any condition for which a MRI procedure is contraindicated.
* Presence of any non-MRI compatible metallic material in the body, such as pacemakers, metallic clips, etc.
* Likelihood of claustrophobia
* Chest circumference greater than that of the helium magnetic resonance (MR) coil.
* Pregnancy, by report of subject. Clinically in the Department of Radiology at UVA, self report is used when screening patients for MR scans as well as CT scans and fluoroscopy studies. If the subject reports there is any chance of their being pregnant a urine pregnancy test will be performed prior to any imaging.

Ages: 4 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yun M Shim, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperpolarized Helium 3 MRI of the Chest
Started | 45
Completed | 44
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hyperpolarized Helium 3 MRI of the Chest
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Ventilation Defects as Seen on Hyperpolarized Helium-3 MRI
Description: On hyperpolarized helium-3 MRI, well ventilated areas of the lung appear bright and poorly ventilated areas appear dark. The poorly ventilated areas are called ventilation defects. Human readers looked at the hyperpolarized helium-3 MR images and determined whether the lungs had: No Defects, Small Defects, or Large Defects.
Time Frame: Day 1
Population: 6 of the 44 imaged subjects were part of the technique development and were not included in the data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperpolarized Helium 3 MRI of the Chest
Number analyzed (Participants) | 38
Participants
  No Defects | 9
  Small Defects | 13
  Large Defects | 16

ADVERSE EVENTS:
Time Frame: 1 week
Description: Patients or their family were contacted within 1 to 5 days after completion of imaging.
Arm/Group | Hyperpolarized Helium 3 MRI of the Chest
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 5/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperpolarized Helium 3 MRI of the Chest (N=44)
Headache/sore throat (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Upset Stomach/vomiting/gas (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT02163681/Prot_SAP_000.pdf